CLINICAL TRIAL: NCT02012153
Title: Autologous Mesenchymal Stromal Cells to Induce Tolerance in Living-donor Kidney Transplant Recipients
Brief Title: Mesenchymal Stromal Cells in Kidney Transplant Recipients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Failure to enroll the number of patients required by the protocol due to the low number of living donor transplants performed at the Clinical Center
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC-Tx tolerance; 2013-003221-29 (EudraCT Number)
Record Dates: First submitted 2013-11-29; First posted 2013-12-16 (Estimated); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Kidney Transplant Rejection
Keywords: Mesenchymal stromal cells; Kidney transplantation; Tolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mesenchymal Stromal Cells (Experimental): A single intravenous infusion of ex-vivo expanded autologous MSCs will be performed in patients in addition to the living-donor kidney transplantation.
  2x10 elevated to sxth power MSCs per kilogram body weight previously isolated from the same recipient will be infused intravenously the day before the kidney transplant procedure.
  Interventions: Biological: Mesenchymal Stromal Cells

INTERVENTIONS:
Biological: Mesenchymal Stromal Cells

SUMMARY:
The general aim of the present study is to test a cell therapy with autologous ex-vivo expanded mesenchymal stromal cells (MSCs) as a strategy to induce tolerance in living-donor kidney transplant recipients. MSCs will be prepared accordingly to established protocols, starting from bone marrow explants of living-donor kidney transplant recipients obtained 3-4 months before kidney transplant. From these samples, MSCs will be expanded in Good Manufacturing Practice (GMP) approved facilities and used for the present study in patients undergoing kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients;
* Aged 18 or older;
* Living-donor (related and unrelated, spouse/husband) kidney transplant recipients;
* Non-Human Leukocyte Antigen (HLA) identical with the donor (one or two haplotype mismatches);
* First kidney transplant;
* Capable of understanding the purpose and risk of the study;
* Written informed consent.

Exclusion Criteria:

* MSC donor positive for HIV-1, HIV-2, hepatitis B virus (HBV),hepatitis C virus (HCV), syphilis;
* Specific contraindication to MSC infusion;
* Any clinical relevant condition that might affect study participation and/or study results;
* Pregnant women and nursing mothers;
* Unwillingness or inability to follow study protocol in the investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-12-04 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
Circulating naïve and memory T cell count (CD45RA/CD45RO) (flow cytometry analysis). | Changes from baseline at 6 and 12 months after transplant.
T-cell function by ELISPOT assay in mixed lymphocyte reaction. | Changes from baseline at 6 and 12 months after transplant.
Number of adverse events. | Changes from baseline up to 48 months.
  At each visit the overall clinical condition of the patient will be evaluated and any adverse event will be recorded.
Circulating regulatory T cell count. | Changes from baseline at 6 and 12 months after transplant.
Urinary FOXP3 mRNA expression evaluated by real time quantitative PCR. | Changes from baseline at 6 and 12 months after transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Study Chair — A.O. Ospedale Papa Giovanni XXIII; Norberto Perico, MD, Study Director — Istituto Di Ricerche Farmacologiche Mario Negri; Giovanni Rota, MD, Principal Investigator — A.O. Ospedale Papa Giovanni XXIII; Federica Casiraghi, Principal Investigator — Istituto Di Ricerche Farmacologiche Mario Negri; Martino Introna, MD, Principal Investigator — Laboratorio G. Lanzani, Bergamo, Italy; Alessandro Rambaldi, MD, Principal Investigator — A.O. Ospedale Papa Giovanni XXIII
Locations (1):
- U.O. Nefrologia e Dialisi, Bergamo, Italy

REFERENCES:
- [Derived] Perico N, Casiraghi F, Todeschini M, Cortinovis M, Gotti E, Portalupi V, Mister M, Gaspari F, Villa A, Fiori S, Introna M, Longhi E, Remuzzi G. Long-Term Clinical and Immunological Profile of Kidney Transplant Patients Given Mesenchymal Stromal Cell Immunotherapy. Front Immunol. 2018 Jun 14;9:1359. doi: 10.3389/fimmu.2018.01359. eCollection 2018. PMID 29963053